CLINICAL TRIAL: NCT01472692
Title: Treatment of Uric Acid With the Xanthine Oxidase Inhibitor Febuxostat: Effects on Blood Pressure, Metabolic Markers, and Aortic Stiffness in Prehypertensive
Brief Title: Study of Febuxostat Effect on Blood Pressure in Patients With High Normal Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 110806
Record Dates: First submitted 2011-11-13; First posted 2011-11-16 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Prehypertension; Gout; Pulse Wave Velocity; Hypertension; 24 Hour Blood Pressure
Keywords: Prehypertension; Gout; Puls Wave Velocity; Hypertension; 24 hour blood pressure
MeSH Terms: conditions — Prehypertension; Gout; Hypertension | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat (Active Comparator)
  Interventions: Drug: Febuxostat
- Placebo (Placebo Comparator)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — 80mg PO daily for 8 weeks
  Other Names: Uloric

SUMMARY:
High normal blood pressure, also called prehypertension, is a significant problem. High uric acid in the blood, the same thing that causes gout, may cause higher blood pressures. The investigators plan to monitor the effects of the drug febuxostat(trade name Uloric) on blood pressure and stiffness of the main blood vessels and see if lowering uric acid has any effect.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertensive male and female subjects with SBP =120-140 mmHg or DBP =80-90 mmHg (as determined by seated office BP).
* Plasma uric acid level ≥5 mg/dl
* Ages 18-50
* non-smokers
* Subjects will need to remain in the San Diego area for the duration of the study and be accessible by telephone or email.

Exclusion Criteria:

* no current smoking in the prior 6 months.
* Any history of any serious medical conditions requiring close monitoring from physicians- such as liver impairment, chronic kidney disease, or diabetes mellitus. Participants not currently under the care of a physician for these conditions will be eligible for the study.
* Any history of gout, hypertension, hypercholesterolemia, morbid obesity.
* Any history of use xanthine oxidase inhibitors, antihypertensives, antiglycemic, and cholesterol lowering medications
* any history of illicit drug use within the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O'Connor, UCSD, Principal Investigator — UCSD; Jason T. Davis, M.D., Study Director — University of California, San Diego
Locations (1):
- Univerisity Of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Gois PHF, Souza ERM. Pharmacotherapy for hyperuricaemia in hypertensive patients. Cochrane Database Syst Rev. 2020 Sep 2;9(9):CD008652. doi: 10.1002/14651858.CD008652.pub4. PMID 32877573

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Principal Investigator for this study has passed away and the results data is not available.
Period: Overall Study
Arm/Group | Febuxostat | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Principal Investigator for this study has passed away and the results data is not available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Changes in 24 Hour Blood Pressure
Time Frame: 8 weeks
Population: The Principal Investigator for this study has passed away and the results data is not available.
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Changes in Pulse Wave Velocity
Time Frame: 8 weeks
Population: The Principal Investigator for this study has passed away and the results data is not available.
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The Principal Investigator for this study has passed away and the results data is not available.
Arm/Group | Febuxostat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The Principal Investigator for this study has passed away and the results data is not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes